CLINICAL TRIAL: NCT00746031
Title: Novel Magnetic Resonance Imaging Strategies as a Non-invasive Biomarker of Vascular and Extracellular Matrix Morphology in Women With Uterine Fibroids.
Brief Title: Novel MRI Strategies as a Non-invasive Biomarker in Women With Uterine Fibroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: PROFESSOR HILARY OD CRITCHLEY, UNIVERSITY OF EDINBURGH
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: REC number 08/MRE00/30
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Fibroid; Leiomyoma
Keywords: MTI; Fibroids; Novel; MR imaging; techniques
MeSH Terms: conditions — Leiomyoma | interventions — Gonadotropin-Releasing Hormone; Goserelin; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): GnRH analogue-Zoladex
  Interventions: Drug: GnRH analogue (Zoladex)
- 2 (Active Comparator): GnRH antagonist plus GnRH analogue
  Interventions: Drug: GnRH analogue (Zoladex); Drug: GnRH antagonist-Cetrorelix
- 3 (No Intervention)

INTERVENTIONS:
Drug: GnRH analogue (Zoladex) — 3.6mg subcutaneous implant. Monthly doses x 3.
  Arms: 1; 2
Drug: GnRH antagonist-Cetrorelix — Subcutaneous injection 3mg x3 over 7 days
  Other Names: Cetrotide
  Arms: 2

SUMMARY:
Fibroids are present in up to 80% of women of reproductive age. Associated heavy menstrual bleeding is often an indication for surgery. At present there are no long-term medical treatments for fibroids. There is an unmet need for a pharmacologic agent able to reduce excessive bleeding and other symptoms associated with increased uterine volume, which could prevent or significantly delay surgery without causing significant unwanted hypoestrogenic side effects and allow preservation of fertility.

The purpose of this study is to investigate and validate novel MR imaging as a non-invasive biomarker for monitoring responses to medical interventions aimed at reduction of excessive menstrual bleeding and decrease in uterine/ fibroid volume. MR imaging is non-invasive, does not involve ionizing radiation and new techniques have the potential to resolve tissue detail to near cellular level.

The investigators are aiming to establish the feasibility and reproducibility of novel MR imaging techniques in the evaluation of treatment response in women with fibroids and to provide mechanistic information on whether the reduction in blood flow of uterine/fibroid vasculature in the shrinkage of fibroids is dependent upon subjects being hypoestrogenic.

ELIGIBILITY:
Inclusion criteria:

* Age>18 years
* Scheduled for hysterectomy with a fibroid uterus
* At least one intramural non-pedunculated, submucosal or subserous fibroid(>2cm) or multiple small fibroids (uterine volume>200cm3)
* Ability to understand and willingness to sign consent form
* Normal smear within 3 years

Exclusion criteria:

* Pregnant or lactating
* Contra indication to MRI
* Unable to tolerate supine position
* Diabetes and/or renal or hepatic impairment
* Contra indication to any of the study medications including gadolinium, MRI contrast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Uterine and fibroid volume | 2010

SECONDARY OUTCOMES:
Uterine vascular perfusion, vasculature and extracellular matrix (ECM)content of fibroids. | 2010

CONTACTS AND LOCATIONS:
Overall Officials: HILARY OD CRITCHLEY, MBChB;MD;FRCOG, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh/ Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Munro KI, Thrippleton MJ, Williams AR, McKillop G, Walker J, Horne AW, Newby DE, Anderson RA, Semple SI, Marshall I, Lewis SC, Millar RP, Bastin ME, Critchley HO. Quantitative serial MRI of the treated fibroid uterus. PLoS One. 2014 Mar 7;9(3):e89809. doi: 10.1371/journal.pone.0089809. eCollection 2014. PMID 24608161